CLINICAL TRIAL: NCT06155864
Title: Imaging Study of Anatomical Variations of the Superficial Temporal Artery
Brief Title: Imaging Study of Anatomical Variations of the Superficial Temporal Artery (EVATSI)
Acronym: EVATSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0119 - EVATSI
Record Dates: First submitted 2023-10-19; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Superficial Temporal Artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: To study the reproducibility of anatomical measurements of the superficial temporal artery using X-ray angio-modensitometry.
- 2: Investigate different CT techniques for studying the superficial temporal artery.
- 3: Study the anatomy of the superficial temporal artery on CT.
- 4: Study the anatomy of the superficial temporal artery on MRI.

SUMMARY:
This study focuses on the anatomy of the superficial temporal artery, an artery of the head. Knowledge of the anatomy of this artery, and the evaluation of methods for exploring it, have implications for clinical medical and surgical practice.

DETAILED DESCRIPTION:
The study will be divided into several parts:

* The aim is to study the reproducibility of anatomical measurements of the superficial temporal artery using CTA.
* The aim is to study the contribution of CTA for the anatomical assessment of the superficial temporal artery.
* The aim is to evaluate the performance of MRI in the anatomical study of the superficial temporal artery.

ELIGIBILITY:
Inclusion Criteria:

* No opposition expressed
* Examination analyzable

Exclusion Criteria:

* Refusal to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent "Polygon of Willis" imaging of the arteries of the head in the medical imaging department of Brest University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Intra- and inter-observer reproducibility of anatomical criteria of the superficial temporal artery in CTA. | 12 months
  The aim is to study the reproducibility of anatomical measurements of the superficial temporal artery. To this end, an intra-class agreement (ICA) analysis will be performed to assess the inter-observer and intra-observer reliability of the measurements. We will also calculate the standard error of measurement (SEM) to assess measurement variability, and perform a Bland-Altman analysis to visualize differences between measurements.
Evaluation of anatomical measurements and reproducibility of measurements obtained with an iterative and classical reconstruction CT technique. | 12 months
  The aim is to compare the performance of the two reconstruction techniques (conventional and iterative) for anatomical assessment of the superficial temporal artery. A repeated-measures analysis of variance can be performed to compare the measurements obtained with the two reconstruction techniques.ICCs and TEMs will also be calculated to assess the reproducibility of measurements with each technique.
Study the anatomy of the superficial temporal artery in a large number of patients, and to correlate the anatomical variants observed with the age of the subjects. | 12 months
  The aim is to study the anatomy of the superficial temporal artery in a large number of patients, and to correlate the anatomical variants observed with the age of the subjects. Descriptive data analysis will be carried out to describe the characteristics of the study population (age, sex, etc.) and the anatomical measurements of the superficial temporal artery.We will use linear regression analysis to assess this relationship and determine the importance of each explanatory variable. We will also assess goodness of fit using measures such as the coefficient of determination R2.
The aim is to compare the performance of arterial time-of-flight (TOF) sequences in MRI at 1.5T and 3T with angio-CT. A comparative analysis of the anatomical measurements obtained with each technique will be carried out. | 12 months
  The aim is to compare the performance of arterial time-of-flight (TOF) sequences in MRI at 1.5T and 3T with angio-CT. A comparative analysis of the anatomical measurements obtained with each technique will be carried out, using t-tests or non-parametric tests depending on the distribution of the data. Concordance between measurements obtained with each technique will be assessed using ICC and Pearson's correlation coefficient.We will seek to identify homogeneous groups of subjects based on their characteristics. We will use cluster analysis to determine the distance between subjects and group them into homogeneous clusters.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifth years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement